CLINICAL TRIAL: NCT00622388
Title: An Open-label, Single-arm. Multi-center Phase 2 Trial With Ofatumumab in Patients With Relapsed/Progressive Diffuse Large B-Cell Lymphoma (DLBCL) Ineligible for Transplant or Relapse/Progression After Autologous Transplant
Brief Title: Ofatumumab in Patients With Relapsed/Progressive Diffused Large B-Cell Lymphoma (DLBCL) Ineligible for or Relapse/Progression After Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111776; GEN415 (Other: Genmab)
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2011-09-08 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-01

CONDITIONS: Lymphoma, Large-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab (Experimental): 8 weekly intra-venous (I.V.) infusions, 1 x 300mg and 7 x 1000mg
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — 8 weekly intra-venous (i.v.) infusions, 1 x 300mg and 7 x 1000mg

SUMMARY:
The purpose of this trial is to determine the effect of ofatumumab in patients with Diffused Large B-Cell Lymphoma (DLBCL) ineligible for transplant or relapsed after autologous transplant

ELIGIBILITY:
Inclusion Criteria:

Patients with DLBCL

* and relapse after complete remission or disease progression after partial remission who are ineligible for autologous stem cell transplantation
* and relapse after complete remission or disease progression after partial remission following autologous stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, London, United Kingdom

REFERENCES:
- [Derived] Coiffier B, Radford J, Bosly A, Martinelli G, Verhoef G, Barca G, Davies A, Decaudin D, Gallop-Evans E, Padmanabhan-Iyer S, Van Eygen K, Wu KL, Gupta IV, Lin TS, Goldstein N, Jewell RC, Winter P, Lisby S; 415 study investigators. A multicentre, phase II trial of ofatumumab monotherapy in relapsed/progressive diffuse large B-cell lymphoma. Br J Haematol. 2013 Nov;163(3):334-42. doi: 10.1111/bjh.12537. Epub 2013 Aug 23. PMID 24032456

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab: Participants received 8 weekly intravenous (iv) infusions of ofatumumab: first infusion of 300 milligrams (mg), followed by 7 infusions of 1000 mg
Period: Overall Study
Arm/Group | Ofatumumab
Started | 81
Completed | 9
Not Completed | 72
Not completed — Disease Progression | 47
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 3
Not completed — Participant Refusal | 1
Not completed — Death | 3
Not completed — Received Alternate Anticancer Therapy | 8
Not completed — Took Prohibited Medication | 2
Not completed — Withdrew Consent | 1
Not completed — Insurance Expired | 1

BASELINE CHARACTERISTICS:
Groups:
- Ofatumumab: Participants received 8 weekly iv infusions of ofatumumab: first infusion of 300 mg, followed by 7 infusions of 1000 mg
Arm/Group | Ofatumumab
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 45
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2
  Hispanic or Latino | 2
  White | 76
  Missing | 1
Number of Participants with the Indicated Prior Therapy [Number; unit: participants] — Study participants had to have either prior autologous stem cell transplant (ASCT) or had to be ineligible for ASCT to be eligible for inclusion.
  participants
    Prior ASCT | 25
    Ineligible for ASCT | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response of ofatumumab treatment was assessed according to the "revised response criteria for malignant lymphoma." Participants with objective response were defined as responders with complete remission (CR) or partial remission (PR) of disease. CR is defined as the disappearance of all evidence of disease, and PR is defined as the regression of measurable disease with no new sites of disease.
Time Frame: 6-month period from start of treatment (up to Week 24)
Population: Full Analysis Set (FAS): all participants who were exposed to study drug irrespective of their compliance to the planned course of treatment
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 81
participants | 9
Statistical Analysis 1: Comparison: Ofatumumab; Test type: Superiority or Other; Response rate = 11, 95% CI 2-sided [5 to 20] — Response rate is calculated as the number of responses divided by the number of participants treated, expressed as a percentage

2. Primary Outcome: Number of Participants Classified as Responders and Non-responders for Objective Response
Description: According to the "revised response criteria for malignant lymphoma," responders included participants with CR and PR, and non-responders included participants with stable disease (SD) and progressive disease (PD). Participants not evaluable (NE) were also considered to be non-responders. PD is defined as any new lesion or an increase by more than or equal to 50% of previously involved sites from baseline. SD is defined as failure to attain CR, PR, or PD.
Time Frame: 6-month period from start of treatment (up to Week 24)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 81
participants
  Responders with CR | 2
  Responders with PR | 7
  Non-responders with SD | 14
  Non-responders with PD | 34
  Non-responders with NE | 24

3. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time from the initial response (CR or PR) to the time of relapse, progression, or death. If the participant was lost to follow-up, the endpoint was censored, and the censoring date was the date of the last attended visit at which the endpoint was assessed.
Time Frame: From date of start of treatment to 2 years or withdrawal
Population: FAS. Only participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab
Number analyzed (Participants) | 9
months | 9.5 [5.4 to NA] — Too few participants experienced the event to estimate the upper limit of the confidence interval.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from treatment start until progression or death.
Time Frame: From date of start of treatment to 2 years or withdrawal
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab
Number analyzed (Participants) | 81
months | 2.5 [2.3 to 4.9]

5. Secondary Outcome: Time to Next Diffuse Large B-Cell Lymphoma (DLBCL) Therapy
Description: Time to next DLBCL therapy was defined as the time from the first infusion date to the time of the first administration of the next DLBCL treatment other than ofatumumab. If the participants were lost to follow-up, the endpoint was censored, and the censoring date was the date of the last attended visit at which the endpoint was assessed.
Time Frame: From date of start of treatment to 5 years or withdrawal
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab
Number analyzed (Participants) | 81
months | NA [7.4 to NA] — Too few participants experienced the event to estimate the median and the upper limit of the confidence interval.

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from first infusion to death. Overall survival was a secondary endpoint in the study. However, since many participants withdrew from the study after developing disease progression overall survival could not be reliably estimated.
Time Frame: From date of start of treatment to 5 years or withdrawal
Population: FAS
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibodies (HAHA) at Screening and at Visits 12, 13, 14, and 18
Description: HAHA are indicators of immune response to ofatumumab. Blood samples were collected from participants at Visits 1, 12, 13, 14, and 18 and analyzed in batches. The number of participants with positive results at each visit is reported.
Time Frame: Screening visit (=<14 days before treatment start), Visit 12 (Month 6), Visit 13 (Month 9), Visit 14 (Month 12), and Visit 18 (Month 24)
Population: FAS. Data are provided for the number of participants attending each visit.
Measure: Number; unit: participants
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 79
participants
  Screening, n=79 | 0
  Visit 12 (Month 6), n=20 | 0
  Visit 13 (Month 9), n=16 | 0
  Visit 14 (Month 12), n=16 | 0
  Visit 18 (Month 24), n=8 | 0
  End of Trial/Withdrawal, n=43 | 0

8. Secondary Outcome: Median Percent Change From Baseline in CD45+CD19+ and CD45+CD20+ Cells in the Peripheral Blood at the Indicated Visits
Description: B cells (CD45+CD19+ and CD45+CD20+) were measured in peripheral blood samples by flow cytometry. Percent change from Baseline = (value at the indicated visits minus the value at Baseline divided by the value at Baseline) * 100.
Time Frame: Baseline and Visit 10 (Week 8), Visit 11 (Week 11), Visit 12 (Month 6), Visit 13 (Month 9), Visit 14 (Month 12), Visit 15 (Month 15), Visit 16 (Month 18), Visit 17 (Month 21), Visit 18 (Month 24), Visit 19 (Month 30), Visit 20 (Month 36)
Population: FAS. Data are provided for the number of participants attending each visit.
Measure: Median (Full Range); unit: percent change in cells
Arm/Group | Ofatumumab
Number analyzed (Participants) | 42
percent change in cells
  CD45+CD19+, Visit 10 (Week 8), n=42 | -100.0 [-100 to 0]
  CD45+CD19+, Visit 11 (Week 11), n=29 | -100.0 [-100 to 56]
  CD45+CD19+, Visit 12 (Month 6), n=18 | -100.0 [-100 to 0]
  CD45+CD19+, Visit 13 (Month 9), n=15 | -100.0 [-100 to 0]
  CD45+CD19+, Visit 14 (Month 12), n=13 | -100.0 [-100 to 0]
  CD45+CD19+, Visit 15 (Month 15), n=12 | -60.7 [-100 to 12]
  CD45+CD19+, Visit 16 (Month 18), n=8 | 6.0 [-88 to 179]
  CD45+CD19+, Visit 17 (Month 21), n=8 | -6.9 [-58 to 56]
  CD45+CD19+, Visit 18 (Month 24), n=7 | -11.1 [-100 to 50]
  CD45+CD19+, Visit 19 (Month 30), n=2 | 80.8 [12 to 150]
  CD45+CD19+, Visit 20 (Month 36), n=2 | 68.6 [-36 to 174]
  CD45+CD20+, Visit 10 (Week 8), n=42 | -100.0 [-100 to 0]
  CD45+CD20+, Visit 11 (Week 11), n=29 | -100.0 [-100 to 56]
  CD45+CD20+, Visit 12 (Month 6), n=18 | -100.0 [-100 to 0]
  CD45+CD20+, Visit 13 (Month 9), n=15 | -100.0 [-100 to 0]
  CD45+CD20+, Visit 14 (Month 12), n=13 | -100 [-100 to 0]
  CD45+CD20+, Visit 15 (Month 15), n=12 | -57.3 [-100 to 0]
  CD45+CD20+, Visit 16 (Month 18), n=8 | 6.0 [-88 to 171]
  CD45+CD20+, Visit 17 (Month 21), n=8 | -6.9 [-58 to 28]
  CD45+CD20+, Visit 18 (Month 24), n=5 | -11.1 [-100 to 50]
  CD45+CD20+, Visit 19 (Month 30), n=2 | 75.2 [7 to 143]
  CD45+CD20+, Visit 20 (Month 36), n=2 | 68.6 [-36 to 174]

9. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. The protocol-defined AE reporting period was from the first infusion (Visit 2/Week 0) to Visit 18 (Month 24 of follow-up) or time of withdrawal (treatment and follow-up).
Time Frame: Time frame is from date of start of treatment to 2 years or withdrawal
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 81
participants | 78

10. Secondary Outcome: Percent Change From Screening in Complement (CH50) Levels
Description: CH50 was mistakenly registered as an outcome measure with the protocol record. Samples were not collected, and no analysis will take place. Thus, no data will be reported for this outcome measure.
Time Frame: Screening and post-baseline visits (last visit was to occur 24 months post first dose)
Population: FAS
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

11. Secondary Outcome: AUC(0-inf) and AUC(0-168) for Ofatumumab at the Eighth Infusion
Description: AUC is defined as the area under the ofatumumab concentration-time curve as a measure of drug exposure. AUC(0-168) is the AUC from the start of infusion to 168 hours after the start of the infusion; AUC(0-inf) is the AUC from the start of infusion extrapolated to infinity.
Time Frame: Visit 9 (Week 7; up to 11 months after last dose)
Population: FAS. Data are provided for the number of participants attending each visit for whom the parameter value could be calculated. Participants contributing AUC(0-inf) data also contributed AUC(0-168) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg.h/mL)
Arm/Group | Ofatumumab
Number analyzed (Participants) | 46
micrograms*hour/milliliter (µg.h/mL)
  AUC(0-inf), n=30 | 720388 (79)
  AUC(0-168), n=46 | 110193 (27)

12. Secondary Outcome: Cmax and Ctrough for Ofatumumab at the First and Eighth Infusions
Description: Cmax is defined as the maximum concentration of drug in serum samples. Ctrough is defined as the minimum observed concentration prior to the start of the next dose. No drug is present prior to the first infusion; therefore, there are no Ctrough results for the first dose.
Time Frame: Visit 2 (Week 0) and Visit 9 (Week 7)
Population: FAS. Data are provided for the number of participants attending each visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 74
micrograms per milliliter (µg/mL)
  First infusion Cmax; 300 mg, n=74 | 109 (42)
  Eighth infusion Cmax; 1000 mg, n=48 | 839 (24)
  Eighth infusion Ctrough; 1000 mg, n=48 | 497 (34)

13. Secondary Outcome: Half-life (T1/2) for Ofatumumab at the Eighth Infusion
Description: t1/2 is defined as terminal half-life and is the time required for the amount of drug in the body to decrease by half.
Time Frame: Visit 9 (Week 7; up to 11 months after last dose)
Population: FAS. Data are provided for the number of participants at each visit for whom the parameter could be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 30
hours | 637 (51)

14. Secondary Outcome: Clearance (CL) of Ofatumumab at the Eighth Infusion
Description: CL is the clearance of drug from serum, which is defined as the volume of serum from which the drug is cleared per unit time.
Time Frame: Visit 9 (Week 7; up to 11 months after last dose)
Population: FAS. Data are presented for the number of participants at each visit for whom the parameter can be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour (mL/h)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 46
milliliters per hour (mL/h) | 9.1 (28)

15. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Ofatumumab at the Eighth Infusion
Description: Vss is the volume of distribution at steady state of ofatumumab.
Time Frame: Visit 9 (Week 7; up to 11 months after the last dose)
Population: FAS. Data are presented for the number of participants attending each visit for whom the parameter can be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Ofatumumab
Number analyzed (Participants) | 30
liters | 8.3 (45)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were reported from first infusion (Week 0) to Month 24 of follow-up (FU)/withdrawal (treatment and FU). Serious AEs were reported through Month 60 (treatment, FU, and extended FU).
Arm/Group | Ofatumumab
Serious Adverse Events (participants affected / at risk) | 33/81
Other Adverse Events (participants affected / at risk) | 68/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=81)
Disease progression (General disorders) | 8
Pyrexia (General disorders) | 2
Infusion related reaction (General disorders) | 1
Multi-organ failure (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Bronchitis (Infections and infestations) | 1
Central line infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neurological symptom (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Eyelid ptosis (Endocrine disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Gastritis (Gastrointestinal disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=81)
Diarrhoea (Gastrointestinal disorders) | 15
Abdominal Pain (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 13
Oedema peripheral (General disorders) | 14
Pyrexia (General disorders) | 9
Asthenia (General disorders) | 6
Disease progression (General disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 12
Anaemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 9
Lymphopenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
Headache (Nervous system disorders) | 5
Blood creatinine increased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 8
Hypersensitivity (Immune system disorders) | 6
Nasopharyngitis (Infections and infestations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.